CLINICAL TRIAL: NCT05187221
Title: Visual, Ocular Surface and Extraocular Diagnostic Criteria for Prevalence of Computer Vision Syndrome: A Cross-sectional Smart-survey Based Study
Brief Title: Prevalence and Sequelae of Computer Vision Syndrome in Egyptian Universities
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Prof. Mohammed Iqbal, Professor of Ophthalmology, Sohag University
Other Study IDs: Soh-Med-21-12-31
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Computer Vision Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control Group: The participants will respond to CVS-F4 questionnaire online via SurveyMonkey to report their potential CVS complains and associated screen factors as screen-time, screen-size, screen-resolution and other factors. This group will contains participants with no CVS complains.
  Interventions: Behavioral: CVS Group

INTERVENTIONS:
Behavioral: CVS Group — CVS-F4 will be an online survey via the SurveyMonkey Company. The participants will report their potential CVS complains and associated screen factors as screen-time, screen-size, screen-resolution and other factors. We will collect the responses and analyse the results. Informed consent will be obtained from the participants as an item within the survey itself that he/she agrees to use his/her data in this research work. This group will contain participants with CVS complains.

SUMMARY:
CVS-F4 questionnaire will be used as an instrument to survey CVS prevalence and severity among medical students

DETAILED DESCRIPTION:
CVS-F4 (30 questions) will be an online survey via the SurveyMonkey Company. We will collect the responses and analyze the results. Informed consent will be obtained from the participants as an item within the survey itself that he/she agrees to use his/her data in this research work. The questionnaire includes questions regarding potential ocular, extra-ocular, musclo-skeletal and neuro-psychatric complains caused by CVS. Complete statistical analysis of the survey data will be done using univariate and multivariate logistic and linear regression analysis. The CVS diagnosis will be based on the 5 diagnostic criteria (5DC) to create a new short self-assessment questionnaire for accurate prevalence of CVS.

ELIGIBILITY:
Inclusion Criteria:

* university students
* university staff members

Exclusion Criteria:

* ocular surgery
* amblyopia
* anisometropia
* strabismus
* systemic disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical students or staff who are using screens in their medical studies or personal lives and how these screens affect their medical studies and the effect of mandated medical computer use if present on their screen-behaviour and associated risk factor
Sampling Method: Probability Sample
Enrollment: 8085 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants suffering from CVS | 3 months
  will be reported in form of percentage (%) of students with CVS
Rate of CVS symptoms-attacks | 3 months
  The results will be presented as annual percentage

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Iqbal, MD, PhD, Principal Investigator — Professor of Ophthalmology
Locations (2):
- Egypt (2):
  - Faculty of medicine, Sohag, Sohag Governorate
  - Faculty of medicine, Sohag

IPD SHARING:
Plan to Share IPD: Yes